CLINICAL TRIAL: NCT05462028
Title: Effectiveness of Vibration Training on Muscle Strength of Lower Limbs, Functional Recovery, and Mood State Among Patients With Acute Stroke
Brief Title: Effectiveness of Vibration Training on Functional Recovery and Mood State Among Patients With Acute Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tri-Service General Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Principal Investigator, CHIA-HUEI LIN, PhD, Associate Professor, Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C202105050
Record Dates: First submitted 2022-07-08; First posted 2022-07-18 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Vibration; Exposure; Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcome data will be collected by a research assistant who was blinded in group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- control group (No Intervention): Only received conventional therapy comprised of standardized treatment and regular rehabilitation (i.e., postural training, facilitation techniques, stretching exercise, and strengthening exercise) prescribed by a rehabilitation physician and performed at 3 to 6 days after admission for five 60-minute sessions per week by the physical, occupational, and speech therapists in the rehabilitation center of the medical center.
- exercise group (Placebo Comparator): The exercise group will receive extra 5 days of 30-minute lower-limb ergometer exercise training in addition to the conventional therapy.
  Interventions: Behavioral: ergometer exercise
- wearable leg vibration training group (Sham Comparator): The wearable leg vibration training group will receive extra 5 days of 30-minute wearable leg vibration of lower limbs combined with 30-minute lower-limb ergometer exercise training at post-vibration session, in addition to the conventional therapy.
  Interventions: Device: Vibration training; Behavioral: ergometer exercise
- lower-extremity weight bearing vibration training group (Experimental): The lower-extremity weight bearing vibration training group will receive extra 5 days of 30-minute lower-extremity weight bearing vibration combined with30-minute lower-limb ergometer exercise training at post-vibration session, in addition to the conventional therapy.
  Interventions: Device: Vibration training; Behavioral: ergometer exercise

INTERVENTIONS:
Device: Vibration training — The vibration sessions were performed and supervised by a stroke care experienced registered nurses/researchers who had both nurse and physiotherapist license. The wearable leg vibration training with vibration frequency = 30 Hz, vibration amplitude = 1 mm in the WG was applied by the wearable leg vibration device (Myovolt, New Zealand) which fits comfortably around the knee and hamstring or calf and delivers focal vibration treatment. While the lower-extremity weight bearing vibration training with vibration frequency = 20 Hz, vibration amplitude = 3 mm in the LG was applied the Cozy Fit (HY-806, China) vibration device with vertical direction, which participants stand with both feet upright on the vibrator in a seated position.
  Arms: lower-extremity weight bearing vibration training group; wearable leg vibration training group
Behavioral: ergometer exercise — ergometer exercise training
  Arms: exercise group; lower-extremity weight bearing vibration training group; wearable leg vibration training group

SUMMARY:
This study aims to exam the effectiveness of vibration training on muscle strength of lower limbs, functional recovery, and mood state among patients with acute stroke.

DETAILED DESCRIPTION:
There remains challenging for improving functional recovery of stroke patients in the acute post-stroke period among patients with acute stroke. Particularly the effectiveness of early rehabilitation combining with vibration training for patients with acute stroke is unknown.

Therefore, this study aims to exam the effectiveness of vibration training on muscle strength of lower limbs, functional recovery, and mood state among patients with acute stroke.

A randomized controlled trial will be conducted. Patients with acute ischemic stroke will be selected and randomly assigned to either control group (CG), exercise group (EG), wearable leg vibration training group (WG), or lower extremity vibration training group (LG). All groups will receive conventional treatment and regular rehabilitation. Neurologic disability (Modified Rankin Scale), muscle strength, functional status (Postural Assessment Scale and Barthel Scale), and mood state (Hospital Anxiety and Depression Scale) will be collected to compare between groups and pre- and post-differences.

ELIGIBILITY:
Inclusion Criteria:

* (1) inpatients diagnosed with acute infarct (ischemic, e.g., large artery atherosclerosis, cardioembolism, and small vessel occlusion) stroke;
* (2) stroke onset occurs within three days of admission;
* (3) aged greater than 20 years and under 80 years;
* (4) able to communicate with verbal or nonverbal methods and understand Mandarin;
* (5) normal cognitive function (Mini-Mental State Examination≥ 21);
* (6) neurologic disability ranged from 1 (able to execute all usual duties and activities despite some symptoms) to 4 (moderately severe , eg., unable to attend to own bodily needs without assistance, and unable to walk unassisted) score evaluated by the modified Rankin Scale (mRS);
* (7) agreed to be randomly assigned

Exclusion Criteria:

* (1) diagnosed with a transient ischemic attack combined with visual and hearing impairment;
* (2) neurologic disability were mRS: 0 (no symptoms) or 5 score (severe disability: requires constant nursing care and attention, bedridden, incontinent) and above;
* (3) an acute/chronic nerve or musculoskeletal injury in lower limbs, or history of bone and joint surgery of low extremities in the past six months;
* (4) a history of cancer, end-stage renal disease with dialysis, dementia, mental health disorders (particularly major depression), based on both of medical records and assessments from the neurologist;
* (5) patients transferred from other wards or intensive care units;
* (6) being unable to participate due to other comorbid neurological and musculoskeletal conditions that produce moderate-to-severe physical disability;
* (7) prolonged stay in hospital for over 21 days due to other medical comorbidities (e.g., myocardial infarction, septic shock, cancer) after admission or length of stay in hospital less than one week due to a decline to treatment and transfer to another hospital for further confirmation of diagnosis and other complementary and alternative therapies.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
neurologic disability | Baseline
  neurologic disability will be assessed by Modified Rankin Scale, which scores are ranged from mRS: 0 (no symptoms) to 6 (death) and score 5 indicates a severe disability: requires constant nursing care and attention, bedridden, and incontinent.
neurologic disability | 5 days after intervention
  neurologic disability will be assessed by Modified Rankin Scale, which scores are ranged from mRS: 0 (no symptoms) to 6 (death) and score 5 indicates a severe disability: requires constant nursing care and attention, bedridden, and incontinent.
neurologic disability | through hospitalization, an average of 14 days
  neurologic disability will be assessed by Modified Rankin Scale, which scores are ranged from mRS: 0 (no symptoms) to 6 (death) and score 5 indicates a severe disability: requires constant nursing care and attention, bedridden, and incontinent.
muscle strength | Baseline
  The reliable and well-validated Medical Research Council Manual Muscle Testing scale, the most commonly accepted method of evaluating muscle strength and easy to perform, will be adopt to evaluate muscle strength. The scale assesses the lower-limb muscle strength of both affected and unaffected side by measuring the resisting gravity load and against the examiner's resistance. The test is scored on a scale of 0 - 5, with 0 indicating the worst muscle strength where no muscle contraction is observed, 1 indicating slight muscle contraction but no limb movement, 2 indicating parallel limb movement but no gravity resistance or lifting, 3 indicating limb movement against gravity, 4 indicating limb movement against slight resistance, and 5 indicating limb movement against moderate resistance.
muscle strength | 5 days after intervention
  The reliable and well-validated Medical Research Council Manual Muscle Testing scale, the most commonly accepted method of evaluating muscle strength and easy to perform, will be adopt to evaluate muscle strength. The scale assesses the lower-limb muscle strength of both affected and unaffected side by measuring the resisting gravity load and against the examiner's resistance. The test is scored on a scale of 0 - 5, with 0 indicating the worst muscle strength where no muscle contraction is observed, 1 indicating slight muscle contraction but no limb movement, 2 indicating parallel limb movement but no gravity resistance or lifting, 3 indicating limb movement against gravity, 4 indicating limb movement against slight resistance, and 5 indicating limb movement against moderate resistance.
muscle strength | through hospitalization, an average of 14 days
  The reliable and well-validated Medical Research Council Manual Muscle Testing scale, the most commonly accepted method of evaluating muscle strength and easy to perform, will be adopt to evaluate muscle strength. The scale assesses the lower-limb muscle strength of both affected and unaffected side by measuring the resisting gravity load and against the examiner's resistance. The test is scored on a scale of 0 - 5, with 0 indicating the worst muscle strength where no muscle contraction is observed, 1 indicating slight muscle contraction but no limb movement, 2 indicating parallel limb movement but no gravity resistance or lifting, 3 indicating limb movement against gravity, 4 indicating limb movement against slight resistance, and 5 indicating limb movement against moderate resistance.
Functional status: Postural Assessment Scale for Stroke | Baseline
  The Postural Assessment Scale for Stroke, consisting of two parts with a 4-point scale and a total score ranging from 0-36, is a well-validated assessment tool for postural control in patients with stroke during the first 3 months after stroke. The PASS will be used to evaluate patient's ability to either maintain posture (including static and dynamic balance) or change posture (switching between lying, sitting, and standing) and participants with higher scores represent a better functional status.
Functional status: Postural Assessment Scale for Stroke | 5 days after intervention
  The Postural Assessment Scale for Stroke, consisting of two parts with a 4-point scale and a total score ranging from 0-36, is a well-validated assessment tool for postural control in patients with stroke during the first 3 months after stroke. The PASS will be used to evaluate patient's ability to either maintain posture (including static and dynamic balance) or change posture (switching between lying, sitting, and standing) and participants with higher scores represent a better functional status.
Functional status: Postural Assessment Scale for Stroke | through hospitalization, an average of 14 days
  The Postural Assessment Scale for Stroke, consisting of two parts with a 4-point scale and a total score ranging from 0-36, is a well-validated assessment tool for postural control in patients with stroke during the first 3 months after stroke. The PASS will be used to evaluate patient's ability to either maintain posture (including static and dynamic balance) or change posture (switching between lying, sitting, and standing) and participants with higher scores represent a better functional status.
Functional status: Barthel Scale | Baseline
  The Barthel Scale, a reliable and well-validated daily life function scale and the most commonly used in long-term care to assess patients' physical functioning, which are highly correlated with the degree of individual disability, will be employed to evaluate the independent daily life function of participants. The scores of the scale with 10 items and several aspects, including eating, movement, personal hygiene, toileting, etc., ranged from 0-100. The higher the score, the better functioning and the more independent in their daily activities the patients have.
Functional status: Barthel Scale | 5 days after intervention
  The Barthel Scale, a reliable and well-validated daily life function scale and the most commonly used in long-term care to assess patients' physical functioning, which are highly correlated with the degree of individual disability, will be employed to evaluate the independent daily life function of participants. The scores of the scale with 10 items and several aspects, including eating, movement, personal hygiene, toileting, etc., ranged from 0-100. The higher the score, the better functioning and the more independent in their daily activities the patients have.
Functional status: Barthel Scale | through hospitalization, an average of 14 days
  The Barthel Scale, a reliable and well-validated daily life function scale and the most commonly used in long-term care to assess patients' physical functioning, which are highly correlated with the degree of individual disability, will be employed to evaluate the independent daily life function of participants. The scores of the scale with 10 items and several aspects, including eating, movement, personal hygiene, toileting, etc., ranged from 0-100. The higher the score, the better functioning and the more independent in their daily activities the patients have.
Mood state | Baseline
  This study will use the Hospital Anxiety and Depression Scale (HADS) to assess the participants' mood state. The reliable and well-validated tool has a total of 14 questions, with seven items related to anxiety (HSDS-A) and seven items related to depression (HADS-D). Each item of the HADS is scored from 0-3, and the total score of both subscales ranged from 0-21. The higher the score, the higher the degree of anxiety or depression of the participants had. A score above 8 indicates the presence of anxiety or depression.
Mood state | 5 days after intervention
  This study will use the Hospital Anxiety and Depression Scale (HADS) to assess the participants' mood state. The reliable and well-validated tool has a total of 14 questions, with seven items related to anxiety (HSDS-A) and seven items related to depression (HADS-D). Each item of the HADS is scored from 0-3, and the total score of both subscales ranged from 0-21. The higher the score, the higher the degree of anxiety or depression of the participants had. A score above 8 indicates the presence of anxiety or depression.
Mood state | through hospitalization, an average of 14 days
  This study will use the Hospital Anxiety and Depression Scale (HADS) to assess the participants' mood state. The reliable and well-validated tool has a total of 14 questions, with seven items related to anxiety (HSDS-A) and seven items related to depression (HADS-D). Each item of the HADS is scored from 0-3, and the total score of both subscales ranged from 0-21. The higher the score, the higher the degree of anxiety or depression of the participants had. A score above 8 indicates the presence of anxiety or depression.

CONTACTS AND LOCATIONS:
Locations (1):
- Chia-Huei Lin, Taipei, Hawaii, Taiwan

IPD SHARING:
Plan to Share IPD: No